CLINICAL TRIAL: NCT04276714
Title: Revofit™ System and Residual Limb Pain in Amputee Patients : Multiple N-of-1 Trial
Brief Title: Revofit™ System Evaluation on Residual Limb Pain in Amputee Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients (difficulty in recruiting according to the inclusion criteria)
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 49RC19_0129
Record Dates: First submitted 2020-02-07; First posted 2020-02-19 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Amputation; Adult Disease
Keywords: residual limbs; pain; adjustable socket
MeSH Terms: conditions — Disease; Pain

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design : multiple N of 1 trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjustable socket (Experimental): First week of the study is with adjustable socket
  Interventions: Other: Socket without Revofit system; Other: Socket with Revofit system
- Classical socket (Experimental): First week of the study is with classical socket
  Interventions: Other: Socket without Revofit system; Other: Socket with Revofit system

INTERVENTIONS:
Other: Socket without Revofit system — All the tests are evaluate during one week with the classical type of fittings
Other: Socket with Revofit system — All the tests are evaluate during one week with the adjustable type of fittings (that is to say with Revofit system)

SUMMARY:
At the early stage of the amputation, the residual limb presents post-surgical fluctuations related to post-operative phase, which would need a frequent prosthetic adjustment. In most cases, the volume of residual limb is constant from 12 to 18 months after surgery. However, some daily fluctuations could appear due to an underlying vascular disease for example, which could be painful and impact the quality of life with a constant need of prosthetics adjustment. The goal of this study is to assess the effectiveness of a system-adjusted fitting in comparison with a standard fitting.

DETAILED DESCRIPTION:
With the " multiple N-of-1 trial " study type, pain, quality of life, functional effects and the patient satisfaction with assistive technology will be assessed for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old and above
* Above knee or below knee amputation (irrespective of etiology and time from amputation)
* Residual limb pain
* Prosthetic with classic fitting
* Fluctuations of residual limb requiring prosthetic adaptation (stump cotton sock, wedgning fitting …)
* Recipients or registered with a social security scheme
* Informed consent form signed beforehand

Exclusion Criteria:

* Patient with peripheral neuropathies contraindicating the use of Revofit system
* Pregnant woman, nursing mother or parturiant
* Patient in detention by judicial or administrative decision
* Patient undergoing psychiatric compulsory care
* Patient in a health or social institution for purposes other than research
* Legally protected person
* Patient unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Pain change assessment | four weeks
  Assess the impact of the Revofit™ system adjusted-fitting on residual limb pain compared to a classic fitting with a daily Visual Analog Scale evaluation [VAS : 0 to 10 which constitues the worst outcome].

SECONDARY OUTCOMES:
Everyday comfort | four weeks
  Quality of life assessed by daily number of adaptation of the prosthesis
Functional effects in twin task | Once a week during four weeks
  A walking analysis by GAITrite once a week
Functional effects in simple task | Once a week during four weeks
  A walking analysis by a six-minute walking distance test once a week
Patient satisfaction with assistive technology | Once a week during four weeks
  Assessment of patient satisfaction by using Quebec User Evaluation of Satisfaction with assistive Technology [QUEST] survey

CONTACTS AND LOCATIONS:
Overall Officials: Mickaël Dinomais, Principal Investigator — MD University hospital Angers; Yoann RONZI, Principal Investigator — MD
Locations (1):
- DIMONAIS, Angers, France

IPD SHARING:
Plan to Share IPD: No